CLINICAL TRIAL: NCT06805123
Title: Comparison of Clinical Outcomes According to Timing of Dietary Restart After Colorectal Endoscopic Submucosal Dissection: A Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Early Feeding Versus Delayed Feeding After Colorectal Endoscopic Submucosal Dissection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Seung Min Hong, Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2411-009-145
Record Dates: First submitted 2025-01-18; First posted 2025-02-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Endoscopic Submucosal Dissection; Colorectal Neoplasms
Keywords: colorectum; endoscopic submucosal dissection; feeding
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: One group undergoes early feeding (< 24 hours), while the other group undergoes late feeding (> 24 hours).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early feeding group (Experimental): The group implementing early feeding (< 24hr).
  Interventions: Other: Early feeding
- Late feeding group (Active Comparator): The group implementing late feeding (> 24hr).
  Interventions: Other: Late feeding

INTERVENTIONS:
Other: Early feeding — Begin drinking water 2 hours after the procedure. If no complications occur 2 hours after starting water intake, progress to a liquid diet. If no abnormalities are observed after the liquid diet, transition to a soft diet for the next meal.
  Arms: Early feeding group
Other: Late feeding — Maintain fasting on the day of the procedure. Begin a liquid diet 24 hours after the procedure. If no complications occur after starting the liquid diet, transition to a soft diet at the next meal.
  Arms: Late feeding group

SUMMARY:
Currently, there are no clear guidelines regarding the optimal timing for dietary restart after gastrointestinal endoscopic submucosal dissection (ESD). While several studies have addressed upper gastrointestinal ESD, a meta-analysis reported that early feeding, initiated within one day after the procedure, showed no statistically significant difference in complication rates compared to delayed feeding initiated after two or more days. Moreover, early feeding was associated with shorter hospital stays and higher patient satisfaction. However, to the best of our knowledge, no studies have investigated early feeding in colorectal ESD.

On the other hand, in the context of surgical procedures involving the gastrointestinal tract, several studies suggest that early feeding may offer clinical advantages over delayed feeding.

The aim of this study is to explore the optimal timing for dietary restart following colorectal ESD. In the early feeding group (<24 hours), patients begin water intake if no abnormalities are observed during a follow-up examination conducted two hours post-procedure. If no further issues arise after an additional two hours, a liquid diet is initiated. In contrast, the delayed feeding group (>24 hours) maintains fasting on the day of the procedure and begins a liquid diet the following day. The study will compare the early and delayed feeding groups in terms of post-ESD early complications (e.g., bleeding, perforation, post-coagulation syndrome), length of hospital stay, patient satisfaction, and delayed complications.

DETAILED DESCRIPTION:
# Sample Size Calculation: This clinical study aims to demonstrate that the experimental group (early feeding group, P1) is not clinically inferior to the control group (delayed feeding group, P2) in patients undergoing colorectal endoscopic submucosal dissection (ESD). The primary efficacy endpoint is set as the incidence rate of early complications within 24 hours post-procedure. For non-inferiority testing, the incidence of early complications (P1 = P2) was assumed to be 3%. The non-inferiority margin (D) was set at 8%, with a significance level (alpha) of 2.5%, power of 80%, and a 1:1 allocation ratio. Using the PASS software (version 11), the calculated sample size was 74 patients per group. Considering a dropout rate of 5%, the required sample size is 78 patients per group, totaling 156 participants.

# Randomization and Blinding: This clinical study employs block randomization to allocate participants to the experimental group (early feeding) and the control group (delayed feeding) in a 1:1 ratio. Blinding will not be applied. A randomization table will be generated independently by a statistician from the Medical Statistics Department of Pusan National University Hospital, using the blockrand package in R (version 4.3.3; R Core Team, 2024, http://cran.r-project.org). The block size will remain blinded.

# Research Participation Procedure: After signing the consent form, the admission process is initiated. Basic tests such as blood tests, ECG, and chest/abdominal X-rays are conducted. Fasting and bowel preparation are performed the day before the procedure.

# Procedure and Initial Management: On the day of the procedure, both groups undergo standard colorectal ESD. Two hours after the procedure, a physical examination, CBC, and chest/abdominal X-rays are performed.

# Dietary Group Classification: Early Feeding Group: If no abnormalities are found during the examination 2 hours after the procedure, water intake begins, followed by a liquid diet and then a porridge diet if no complications occur.

Late Feeding Group: Patients remain fasting on the day of the procedure. A liquid diet begins 24 hours after the procedure, followed by a porridge diet if no complications occur.

# Survey: Patient satisfaction is evaluated through a survey. Patients visit the outpatient clinic after discharge to review procedural outcomes and assess for delayed complications.

# Observation Items: Age, sex, height, weight, BMI, underlying diseases (hypertension, diabetes, cerebrovascular disease, ischemic heart disease, other heart diseases, atrial fibrillation (or atrial flutter), other arrhythmias, chronic kidney disease, dialysis status, liver cirrhosis, other vascular diseases), history of previous abdominal surgery, smoking history, alcohol consumption history, medication history (aspirin, clopidogrel, other antithrombotic agents, warfarin, direct oral anticoagulants (DOACs), nonsteroidal anti-inflammatory drugs (NSAIDs), steroids), type of bowel preparation used, pre-procedure serum white blood cell count, pre-procedure serum hemoglobin, pre-procedure serum platelet count, pre-procedure absolute neutrophil count, pre-procedure prothrombin time (PT) (including INR), pre-procedure activated partial thromboplastin time (aPTT), post-procedure serum white blood cell count, post-procedure serum hemoglobin, post-procedure serum platelet count, post-procedure absolute neutrophil count, location of the lesion, size of the lesion (long axis, short axis), macroscopic morphology of the lesion, degree of submucosal fibrosis, resection method, resection time, post-resection management time, total procedure time, type of post-resection management performed, en bloc resection status, occurrence of complications during the procedure, measures taken for intra-procedural complications and their outcomes, occurrence of complications within 24 hours post-procedure, measures taken for complications within 24 hours post-procedure and their outcomes, occurrence of complications beyond 24 hours post-procedure, measures taken for complications beyond 24 hours post-procedure and their outcomes, length of hospital stay (days), pathology results (histology, differentiation grade, invasion depth, horizontal resection margin, vertical resection margin, lymphatic invasion, vascular invasion, perineural invasion), number of days until outpatient follow-up after discharge, patient satisfaction (Likert scale).

# Data Analysis and Statistical Methods: Descriptive statistics will be used to summarize the data: continuous variables will be presented as the number of observations, mean, standard deviation, minimum, maximum, and quartiles, while categorical variables will be presented as frequencies and percentages. Group comparisons will be conducted using an independent t-test or Wilcoxon rank-sum test for continuous variables and a chi-square test or Fisher's exact test for categorical variables. To confirm the non-inferiority of the treatment group (T) compared to the control group (C), the two-sided 95% confidence interval for the difference in proportions (T-C) will be calculated. Non-inferiority will be established if the upper limit of the confidence interval is within the predefined non-inferiority margin. A two-sided test will be performed at a significance level of 5%. No interim analysis will be conducted in this clinical study, and no imputation methods for missing data will be applied.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing colorectal endoscopic submucosal dissection for the following lesions:

* Differentiated early colorectal cancer confined to the mucosa, without ulcers, and measuring ≤5 cm
* Laterally spreading tumors measuring ≥2 cm
* Sessile polyps measuring ≥2 cm
* Adenomas accompanied by fibrosis
* Differentiated early cancer of the colon or rectum without lymph node metastasis, aside from those covered by partial self-payment insurance (Korean National Health insurance)
* Submucosal tumors of the colon or rectum
* Patients who have signed the consent form to participate in this study

Exclusion Criteria:

* Under 18 years of age
* Patients with unresolved colorectal cancer
* Patients with non-remissive inflammatory bowel disease (IBD)
* Patients with blood coagulation disorders
* Patients with a prothrombin time (PT) INR ≥ 1.5 despite medical correction
* Pregnant patients
* Patients who refuse to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Complication | Through study completion, an average of 1 year
  Bleeding, perforation, Post procedural coagulation syndrome

SECONDARY OUTCOMES:
Length of hospital stay | through study completion, an average of 1 year
  The number of days from admission to discharge
patient satisfaction | through study completion, an average of 1 year
  Patient satisfaction is assessed through a survey conducted with the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Dong Hoon Baek, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (5):
- South Korea (5):
  - Inje university busan paik hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin university gospel hospital, Busan
  - Ulsan university hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sang Un Park, Dong Kyung Chang. Endoscopic Submucosal Dissection for Colorectal Tumors. Korean J Gastrointest Endosc 2010;40.
- [Background] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Background] Hirao M, Masuda K, Asanuma T, Naka H, Noda K, Matsuura K, Yamaguchi O, Ueda N. Endoscopic resection of early gastric cancer and other tumors with local injection of hypertonic saline-epinephrine. Gastrointest Endosc. 1988 May-Jun;34(3):264-9. doi: 10.1016/s0016-5107(88)71327-9. No abstract available. PMID 3391382
- [Background] Gotoda T, Kondo H, Ono H, Saito Y, Yamaguchi H, Saito D, Yokota T. A new endoscopic mucosal resection procedure using an insulation-tipped electrosurgical knife for rectal flat lesions: report of two cases. Gastrointest Endosc. 1999 Oct;50(4):560-3. doi: 10.1016/s0016-5107(99)70084-2. No abstract available. PMID 10502182
- [Background] Hosokawa K, Yoshida S. [Recent advances in endoscopic mucosal resection for early gastric cancer]. Gan To Kagaku Ryoho. 1998 Mar;25(4):476-83. Japanese. PMID 9530352
- [Background] Ono H, Kondo H, Gotoda T, Shirao K, Yamaguchi H, Saito D, Hosokawa K, Shimoda T, Yoshida S. Endoscopic mucosal resection for treatment of early gastric cancer. Gut. 2001 Feb;48(2):225-9. doi: 10.1136/gut.48.2.225. PMID 11156645
- [Background] Masakatsu Fukuzawa, Takuji Gotoda. History of endoscopic submucosal dissection and role for colorectal endoscopic submucosal dissection: A Japanese perspective. Gastrointestinal Intervention 2012;1:30-35.
- [Background] Tanaka S, Terasaki M, Kanao H, Oka S, Chayama K. Current status and future perspectives of endoscopic submucosal dissection for colorectal tumors. Dig Endosc. 2012 May;24 Suppl 1:73-9. doi: 10.1111/j.1443-1661.2012.01252.x. PMID 22533757
- [Background] Kim ER, Chang DK. Management of Complications of Colorectal Submucosal Dissection. Clin Endosc. 2019 Mar;52(2):114-119. doi: 10.5946/ce.2019.063. Epub 2019 Mar 29. PMID 30959586
- [Background] Watanabe J, Watanabe J, Kotani K. Early vs. Delayed Feeding after Endoscopic Submucosal Dissection for Gastric Cancer: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2020 Nov 27;56(12):653. doi: 10.3390/medicina56120653. PMID 33261059
- [Background] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale RG, Waitzberg D, Bischoff SC, Singer P. ESPEN practical guideline: Clinical nutrition in surgery. Clin Nutr. 2021 Jul;40(7):4745-4761. doi: 10.1016/j.clnu.2021.03.031. Epub 2021 Apr 19. PMID 34242915
- [Background] Canzan F, Longhini J, Caliaro A, Cavada ML, Mezzalira E, Paiella S, Ambrosi E. The effect of early oral postoperative feeding on the recovery of intestinal motility after gastrointestinal surgery: a systematic review and meta-analysis of randomized clinical trials. Front Nutr. 2024 May 16;11:1369141. doi: 10.3389/fnut.2024.1369141. eCollection 2024. PMID 38818132
- See also: Ministry for Health, Welfare and Family Affairs, National Cancer Center. National cancer information center — http://www.cancer.go.kr/cms/statics/incidence/index.html